CLINICAL TRIAL: NCT06525194
Title: An Interprofessional Education Program Based on the ARCS-V Motivation Model on the Theme of "Chronic Disease Management and Patient Safety": An Action Research
Brief Title: An Interprofessional Education Program
Acronym: ARCS-V
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Aysel Başer, assistant professor dr, Izmir Democracy University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MedEdu1
Record Dates: First submitted 2024-07-19; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Education; Professional Role; Interprofessional Relations; Patient Safety; Acceptability of Health Care; Patient Acceptance of Health Care
Keywords: Interprofessional Education; ARCS_V Motivational Model; Medical Education; Health Professionals; Action Research; ADDIE Insctructional Design
MeSH Terms: conditions — Patient Acceptance of Health Care | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The program was based on the ARCS-V motivational design model, included three sessions and was hybrid.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational Intervention Group (Experimental): Participants in this group included undergraduate healthcare students from the faculties of dentistry, medicine, and health sciences at a higher education institution in Turkey. The group underwent an interprofessional education (IPE) program designed based on the ARCS-V motivational design model. The program consisted of three sessions and was delivered in a hybrid format, incorporating both online and face-to-face elements. Various tactics and strategies from the motivational model were used throughout the training process. The Readiness for Interprofessional Learning Scale (RIPLS) and the ARCS-V Motivation Scale were administered to assess the students' readiness for interprofessional education and the program's effectiveness. The educational content included scenarios, multimedia elements, messages, emails, reflection assignments, and group tasks, which aimed to enhance students' motivation, interest, and overall learning experience.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — An Interprofessional Education Program Based on the ARCS-V Motivation Model on the Theme of "Chronic Disease Management and Patient Safety"

SUMMARY:
Aim: The aim of the study was to develop and implement an interprofessional education (IPE) program that will enhance healthcare students' learning through motivating them with a theme. Methods: Undergraduate healthcare students enrolled in faculties of dentistry, medicine, and health sciences at a higher education institution in Turkey participated in this program. The program was based on the ARCS-V motivational design model, included three sessions and was hybrid. Tactics and strategies from the motivational model were used throughout the online and face-to-face training process. The Readiness for Interprofessional Learning Scale (RIPLS) was used to assess students' readiness for interprofessional education, while the ARCS-V Motivation Scale was used to assess the program. Data were analyzed using Chi-Square test, Independent t test, Wilcoxon rank test, Mann Whitney U test, and one way analysis of variance.

DETAILED DESCRIPTION:
The IPE program titled Chronic Disease Management and Patient Safety was carried out as a hybrid (online and face-to-face) and three-session program with a focus on interprofessional communication. The program provided students interprofessional collaboration, communication, roles and responsibilities, ethics, lifelong learning, and health service delivery skills based on patient needs and teamwork.

For this program, an announcement was made through the faculties which provide healthcare education and volunteering students from the Faculties of Dentistry, Medicine and Health Sciences (Nutrition and Dietetics, Nursing, Physical Therapy and Rehabilitation) were included in the education program. A whatsapp group of volunteer students was created and used for communication and motivational strategies. The link was sent to the students ahead of time via e-mail and the whatsapp group. The tactics and strategies required by the ARCS-V Motivation Model were used throughout the whole process.

• First session: In this session, which was online and lasted for 120 minutes, the education program was introduced to the students and conceptual information was presented. Links to the sociodemographic data form and the RIPLS were shared with the students and they were asked to fill them out prior to face to-face training.

The second and third sessions were face-to-face and were comprised of two 8-hour work days. Facilitators and students participated in these sessions.

• Second session: Introductions and warm-up exercises were carried out. In the development phase of the ADDIE instructional design, four scenarios addressing "Chronic Disease Management and Patient Safety" which involved different health professionals were prepared. The participants were segmented into four study groups, each delineated by their respective professional domains.The formation of these groups was intentionally designed to include a proportional mix of professional fields relevant to each specific scenario. For example, the makeup of one scenario group included 2 medical students, 2 nursing students, 1 physiotherapy student, and 2 dentistry students. In a parallel manner, a different scenario group was arranged with 2 students from medicine, 2 from nursing, 1 from dentistry, and 2 focusing on nutrition and dietetics. This strategic grouping fostered a diverse yet balanced professional composition in each group, directly aligning with the scenario-driven learning objectives.

Two facilitators and one observer were appointed to each group. The task of the facilitators was to ensure that the scenario was read by the students and the discussion was guided by discussion questions.

Observers watched the students and facilitators and took notes on the process of conducting the guided discussion as part of the interprofessional education program.

The whole discussion process was audio- and video-recorded with the voluntary consent of the students and facilitators.

At the end of the day;

* Each group was asked to make a presentation of their achievements according to the interprofessional education competencies (roles and responsibilities, communication skills, collaborative leadership, teamwork, ethics, approach to patient needs and lifelong learning) in the scenarios they discussed.
* Each student was scored by the facilitators using the IPE evaluation form.
* Each student was given questions prepared for reflection based on the scenario they discussed and asked to submit them to the facilitators as homework within a few hours.
* In preparation for the next day, all facilitators were provided with the discussion session recordings and students' reflection assignments and were asked to prepare feedback.

  * Third Session: This session was planned in a large group format including students, facilitators, and observers.

The session started with a warm-up chat. A presentation on the outcomes of the discussion were made by the student who had the role of spokesperson in each group.

The facilitators showed the discussion video segments to the whole group and gave feedback by sharing the positive ideas and the ideas that needed to be improved. They presented the content analysis of the student reflection assignments.

At the end of the session, verbal feedback was received from all participants regarding the implementation. Certificates were given to all participants.

The ARCS-V motivation model scales and the RIPLS were administered to the students.

ELIGIBILITY:
Inclusion Criteria:

* To be a health professional student at the undergraduate level in the Faculty of Dentistry, Medicine and Health Sciences (Nutrition and Dietetics, Nursing, Physical Therapy and Rehabilitation) at Izmir Democracy University in Turkey.
* Voluntarily participate in the training.

Exclusion Criteria:

* Being a student at universities other than Izmir Democracy University

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-07-02 (Actual); Primary Completion 2022-07-02 (Actual); Study Completion 2022-07-03 (Actual)

PRIMARY OUTCOMES:
The Readiness for Interprofessional Learning Scale (RIPLS) | 2 days
  The Readiness for Interprofessional Learning Scale (RIPLS) was developed by Parsell and Bligh (1999), revised by McFadyen et al. (2005,2009) and adapted to Turkish by Ergönül et al. This scale is a three-dimensional, five-point Likert type scale consisting of 19 items used to measure participants' attitudes towards teamwork and collaboration, professional identity, and roles and responsibilities. According to the literature, a score of 4 and above indicates increased readiness.
ARCS-V Motivation Scale | 2 days
  The study utilized the ARCS-V motivation model alongside the ADDIE instructional design model. ARCS-V Motivation Design Scales, 5-point Likert type scales where higher scores indicate higher motivation, assessed the effectiveness of motivational strategies in the IPE program.
  Scales Used:
  Instructional Materials Motivation Survey (IMMS): Developed by Keller in 1993 and revised in 2009, this scale has 16 items focusing on attention, relevance, confidence, and satisfaction.
  Course Interest Survey (CIS): Created by Keller in 1993, it also consists of 16 items, targeting the same four factors as IMMS.
  Volition For Learning Scale (VFLS): Developed by Keller et al. in 2020, this 13-item scale is two-dimensional, focusing on action planning and action control, reflecting the need for motivation, volition, and self-regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Baser, Asst Prof, Principal Investigator — Izmir Democracy University
Locations (1):
- İzmir Demokrasi Üniversitesi Tıp Fakültesi, Izmir, Konak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No